CLINICAL TRIAL: NCT05263232
Title: Natural Daylight to Improve 24h Metabolism and Glucose Control in Type 2 Diabetes
Brief Title: Metabolic Effects of Natural Office Light in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Velux Fonden (Other); University of Geneva, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL77984.068.21
Record Dates: First submitted 2022-01-07; First posted 2022-03-02 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2; Circadian Dysregulation
Keywords: circadian rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronobiology Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural office light (Experimental): Over 4.5 days, participants will stay inside in an office room from 8:00 to 17:00h with wide transparent windows under natural daylight.
  Interventions: Other: Natural or artificial office light exposure
- Artificial office light (Experimental): Over 4.5 days, participants will stay inside in an office room from 8:00 to 17:00h with shielded windows under artificial light.
  Interventions: Other: Natural or artificial office light exposure

INTERVENTIONS:
Other: Natural or artificial office light exposure — Over 4.5 days, participants will stay at our research facilities under different light conditions. Over these days different measurements will take place, including 24h continuous glucose monitoring, 24h blood and saliva sampling, 24h blood pressure and heart rate assessments, 24h core and skin temperature assessments, 24h energy expenditure and whole-body substrate metabolism, and a skeletal muscle biopsy and a mixed meal tolerance test with indirect calorimetry will be performed on the respectively last test day.

SUMMARY:
This study will investigate the potential benefit of scheduled natural daylight exposure to improve glucose control in type 2 diabetes (T2D) patients and to unravel molecular mechanisms underlying the effects of natural daylight on circadian clocks and (glucose) metabolism in human skeletal muscle from T2D patients. Participants will stay at our research facilities and will be exposed to natural daylight or artificial light during the daytime over 4.5 days in a randomized cross-over design. For both conditions, the evening and night will be spent under standardized dim and dark conditions.

DETAILED DESCRIPTION:
Obesity and type 2 diabetes (T2D) are both strongly associated with a westernized lifestyle of low physical activity levels and high caloric intake. However, recently it has been recognized that also our 24-hour culture, characterized by working and eating late, reduced sleep (quantity and quality), and excessive light exposure in the evening and at night, should be considered as lifestyle factors that may negatively impact metabolic health. In this context, a factor that is often overlooked and underestimated is the lack of natural daylight since most people spend almost their entire work time in indoor office environments with limited access to natural daylight through windows.

Therefore, this study investigates the potential benefit of scheduled natural daylight exposure to improve glucose control in T2D individuals and to unravel molecular mechanisms underlying effects of natural daylight on circadian clocks and (glucose) metabolism in human skeletal muscle from T2D patients. For this purpose, overweight to obese T2D patients (male and female) will undergo a randomized cross-over trial in which each subject serves as its own control. Participants will stay at our research facilities and will be exposed to natural daylight or artificial light during the daytime over 4.5 days. For both conditions, the evening and night will be spent under standardized dim and dark conditions, respectively. Over these two 4.5 days intervention periods, extensive 24h metabolic profiling will be conducted, including 24h continuous glucose monitoring, 24h blood and saliva sampling, 24h blood pressure and heart rate assessments, 24h core and skin temperature assessments, 24h energy expenditure and whole-body substrate metabolism, and a skeletal muscle biopsy and a mixed meal tolerance test with indirect calorimetry will be performed on the respectively last test day.

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to provide signed and dates written consent prior to any study specific procedures
* Male + females (postmenopausal defined as at least 1 year post cessation of menses)
* T2DM duration at least 1 year
* BMI: ≥ 25 kg/m²
* Age: 40-75
* Well-controlled diabetes with respect to glycemic control and on stable anti-diabetes medication regimes
* Habitual bedtime of 23:00 ± 2h
* Regular sleep duration (7-9 h/night)
* Stable dietary habits: no weight gain or loss > 5 kg in the last three months

Exclusion Criteria:

* Insulin treatment
* Uncontrolled hypertension
* Signs of active diabetes-related co-morbidities like active cardiovascular diseases, active diabetic foot, polyneuropathy or retinopathy
* Signs of active liver or kidney malfunction
* Use of SGLT2 inhibitors
* Using > 400mg caffeine daily (more than 4 coffee or energy drink)
* Extreme early bird or extreme night person (score ≤30 or ≥70 on MEQ-SA questionnaire)
* shift work or travel across more than one time zone in the 3 months before the study
* Heavily varying sleep-wake rhythm
* Frequent engagement in programmed exercise as judged by the investigator
* Any medication that will interfere with the study outcomes or hamper the safety of the participant
* Alcohol consumption of >2 servings per day for men and >1 serving per day for woman
* Significant food allergies/intolerance (seriously hampering study meals)
* Subjects who do not want to be informed about unexpected medical findings during the screening /study, or do not wish that their physician is informed
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the Investigator
* Smoking in the past 6 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
average 24h blood glucose levels | continously over 4.5 days
  Interstistial glucose levels determined by continuous glucose monitoring

SECONDARY OUTCOMES:
Postprandial metabolism upon a mixed-meal tolerance test (energy expenditure) | measured at 9:00, 9:30, 10:00, 11:00, 12:00 and 13:00 on Day 5
  Energy expenditure (kJ/min) measured by indirect calorimetry
Postprandial metabolism upon a mixed-meal tolerance test (carbohydrate oxidation) | measured at 9:00, 9:30, 10:00, 11:00, 12:00 and 13:00 on Day 5
  Carbohydrate oxidation (μmol/kg x min) measured by indirect calorimetry
Postprandial metabolism upon a mixed-meal tolerance test (fatty acid oxidation) | measured at 9:00, 9:30, 10:00, 11:00, 12:00 and 13:00 on Day 5
  Fatty acid oxidation (μmol/kg x min) measured by indirect calorimetry
Postprandial plasma metabolites upon a mixed-meal tolerance test (glucose) | measured at 9:00, 9:15, 9:30, 9:45, 10:00, 10:30, 11:00, 11:30, 12:00, 13:00 on Day 5
  Plasma glucose levels determined from venous blood draws
Postprandial plasma metabolites upon a mixed-meal tolerance test (insulin) | measured at 9:00, 9:15, 9:30, 9:45, 10:00, 10:30, 11:00, 11:30, 12:00, 13:00 on Day 5
  Plasma insulin levels determined from venous blood draws
Postprandial plasma metabolites upon a mixed-meal tolerance test (free fatty acids) | measured at 9:00, 9:15, 9:30, 9:45, 10:00, 10:30, 11:00, 11:30, 12:00, 13:00 on Day 5
  Plasma FFA levels determined from venous blood draws
Postprandial plasma metabolites upon a mixed-meal tolerance test (triglycerides) | measured at 9:00, 9:15, 9:30, 9:45, 10:00, 10:30, 11:00, 11:30, 12:00, 13:00 on Day 5
  Plasma triglyceride levels determined from venous blood draws
Skeletal muscle biopsy outcomes (Circadian transciptome) | muscle tissue taken at 7:30h on Day 5
  Quantify DNA by micro-array
Culturing human primary myotubes to assess circadian reporter characteristics | muscle tissue taken at 7:30h on Day 5
  in vivo culturing of primary myotubes

OTHER OUTCOMES:
24 hour energy expenditure | measured at 8:00, 13:00, 18:00 and 22:30 on Day 4
  Energy expenditure (kJ/min)
24h whole-body energy metabolism (cabrohydrate oxidation) | measured at 8:00, 13:00, 18:00 and 22:30 on Day 4
  Carbohydrate oxidation (μmol/kg x min) measured by indirect calorimetry
24h whole-body energy metabolism (fatty acid oxidation) | measured at 8:00, 13:00, 18:00 and 22:30 on Day 4
  Fatty acid oxidation (μmol/kg x min) measured by indirect calorimetry
24h profiles of plasma metabolites (i.e. free fatty acids, triglycerides, insulin) | measured on Day 4 at 8:00, 10:00, 12:00, 13:00, 14:00, 16:00, 18:00, 20:00, 22:00, 23:00, and on Day 5 at 00:00, 02:00, 04:00 and 06:00h
  Plasma levels determined from venous blood draws
Mass spectrometry-based 24h serum lipidomics | measured on Day 4 at 8:00, 12:00, 16:00, 20:00, and on Day 5 at 00:00, 04:00 and 8:00
  analysis of all lipid species evident in serum
Sleep quality questionnaire (Leeds Sleep Evaluations Questionnaire - LSEQ) | after each of the 4 nights
  LSEQ scores
Sleep quality questionnaire (Pittsburgh Sleep Quality Index - PSQI) | after each of the 4 nights
  PSQI scores
24h blood pressure | measured hourly from 7:00 to 23:00h on Day 4, and every second hour from 0:00 to 6:00 on Day 5
  blood pressure (mmHg)
24h heart rate | measured continously over 4.5 days
  heart rate (bpm) assesses through chest-worn heart rate monitor
24h skin temperature | measured continously on Day 3
  skin temperature (°C) assessed via wireless temperature sensors (iButtons)
24h core body temperature | measured continously on Day 3
  Core body temperature measured by an ingested telemetric pill (°C)
mRNA in peripheral blood mononuclear cells (PBMC) of markers involved in the molecular clock | blood samples taken on Day 4 at 8:00, 13:00, 18:00, 23:00, and on Day 5 at 4:00 and 9:00
  Quantify mRNA levels by micro array

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided